CLINICAL TRIAL: NCT01350115
Title: A Phase II, Double-blind, Randomized, Proof-of-Concept, Dose-ranging Trial Evaluating the Efficacy, Safety and Pharmacokinetics of Oral LDE225 in Treatment of Adult Patients With Nevoid Basal Cell Carcinoma Syndrome
Brief Title: Efficacy, Safety and Pharmacokinetics of Oral LDE225 in Treatment of Patients With Nevoid Basal Cell Carcinoma Syndrome (NBCCS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLDE225B2209; 2010-023819-34 (EudraCT Number)
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Basal Cell Carcinoma; Gorlin Syndrome; Nevoid Basal Cell Carcinoma Syndrome
Keywords: Basal Cell Carcinoma; Gorlin Syndrome,; Gorlin-Goltz Syndrome,; Basal Cell Nevus Syndrome,; Nevoid Basal Cell Carcinoma Syndrome,; Basal Cell Carcinoma Nevus Syndrome; Smo inhibitor,; Hedgehog pathway inhibitor; BCCs
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — sonidegib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDE225 (Active Comparator): Participants received 400 mg once daily.
  Interventions: Drug: LDE225
- Placebo (Placebo Comparator): Participants received matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LDE225 — supplied as 100 mg capsules
  Arms: LDE225
Drug: Placebo — supplied in capsules
  Arms: Placebo

SUMMARY:
This was a phase II, double-blind, randomized, proof-of-concept, dose-ranging trial evaluating the efficacy, safety and pharmacokinetics of oral LDE225 in treatment of adult patients with NBCCS. This was an exploratory study designed to demonstrate preliminary efficacy of LDE225 in this indication. This study included a Screening period of approximately 4 weeks, treatment period duration of 12 weeks with initial follow-up of approximately 6-8 weeks followed by a long-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple basal cell carcinomas (at least two) and typical presentation of NBCCS.
* Female patients must be women of non-childbearing potential (WONCBP).

Exclusion Criteria:

* Use of any topical treatment to treat BCCs, including prescription and over the counter in the 4 weeks prior to first dose of study drug.
* Use of photodynamic therapy (PDT), radiation or systemic treatment known to affect BCCs or neoplasm in the 12 weeks prior to first dose of study drug.
* Patients receiving medications that are recognized to cause rhabdomyolysis or patients with a prior history of rhabdomyolysis.
* Patients with a histologically confirmed diagnosis of locally advanced or metastatic BCC.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Leuven, Belgium
- Canada (3):
  - Novartis Investigative Site, Markham, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Kiel, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to one of the following 2 treatment arms in a ratio of 6:1,LDE225 400 mg QD and Placebo QD.
Period: Core Study (All Patients)
Arm/Group | LDE225 | Placebo
Started | 8 | 2
Safety Anlysis Set | 8 | 2
Pharmacodynamic Set | 7 | 2
Completed | 8 | 2
Not Completed | 0 | 0
Period: Long Term Follow-Up (All Patients)
Arm/Group | LDE225 | Placebo
Started | 8 | 2
Completed | 7 | 0
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDE225 | Placebo | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (9.90) [37 to 68] | 66 (2.00) [64 to 68] | 53.6 (10.95) [37 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Clearance Assessment of Main Target Basal Cell Carcinomas (BCCs)
Description: The clinical response of the main target (and secondary target, as appropriate) BCC(s) to treatment was evaluated using the following 6-point scale comparing the assessment at the visit to the clinical presentation at Baseline: 0 = Worsening, 1 = No change, 2 = Slight clearance (1-25% improvement), 3 = Moderate clearance (26-75% improvement), 4 = Marked clearance (76-99% improvement),5 = Complete clearance (100% improvement) Complete clearance was defined as no clinical residual signs of carcinoma, as evaluated by the Investigator at a post-Baseline visit, with the exception of post-inflammatory changes such as minimal residual erythema or residual hyper-pigmentation or hypo-pigmentation or residual scarring.
Time Frame: Day 113
Population: All participants, who had evaluable (or complete) pharmacodynamic (PD) or biomarker parameter data and were without protocol deviations with significant impact on the PD data, were included in the PD analysis set.
Measure: Number; unit: Participants
Arm/Group | LDE225 | Placebo
Number analyzed (Participants) | 7 | 2
Participants
  Complete Clearance (100% Improvement) | 3 | 0
  Marked Clearance (76-99% Improvement) | 3 | 0
  Moderate Clearance (26-75% improvement) | 1 | 0
  Slight Clearance (1-25%) | 0 | 1
  Worsening | 0 | 1

2. Secondary Outcome: Histological Clearance Assessment of Main Target BCCs
Description: The main (and secondary, if appropriate) target BCC tumor area(s) was/were excised surgically and sent to a central laboratory for histological examination.
Time Frame: day 113
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | LDE225 | Placebo
Number analyzed (Participants) | 7 | 2
Percentage of participants
  Histological clearance | 57 | 0
  Complete clinical (up to day 85) & histological | 14 | 0
  Complete clinical (up to day 113) & histological | 29 | 0

3. Secondary Outcome: Measure: Disease Burden by BCC Tumor Counts
Description: BCC tumor counts were performed separately for five body regions: head and neck, trunk back, trunk front (including axillae and groin), upper extremities and lower extremities (including buttocks). During the counting, the BCC tumors, were categorized upon inspection by their longest diameter measurement (<10 mm, 10-19 mm, 20-29 mm, and >+30mm), and also by the type of BCC (superficial, nodular, other). The counts for all of the BCC type and size categories were determined (or estimated if many small lesions) for each body region. The body region counts were summated to provide the overall BCC tumor count.
Time Frame: Baseline, day 85, and day 113
Population: as for outcome 1
Measure: Number; unit: Number of BCC tumors
Arm/Group | LDE225 | Placebo
Number analyzed (Participants) | 7 | 2
Number of BCC tumors
  Baseline | 566 | 510
  Day 85 | 341 | 571
  Day 113 | 309 | 619

ADVERSE EVENTS:
Groups:
- LDE225 - Core: Participants received 400 mg once daily.
- Placebo - Core: Participants received matching placebo.
Arm/Group | LDE225 - Core | Placebo - Core | LDE225 - Long Term Follow-up | Placebo - Long Term Follow-up
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/2 | 1/8 | 0/2
Other Adverse Events (participants affected / at risk) | 7/8 | 1/2 | 2/8 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 - Core (N=8) | Placebo - Core (N=2) | LDE225 - Long Term Follow-up (N=8) | Placebo - Long Term Follow-up (N=2)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 - Core (N=8) | Placebo - Core (N=2) | LDE225 - Long Term Follow-up (N=8) | Placebo - Long Term Follow-up (N=2)
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.